CLINICAL TRIAL: NCT01091051
Title: Safety and Efficacy of Ustekinumab in the Treatment of Patients With Palmo-Plantar Pustular Psoriasis or With Palmo-Plantar Pustulosis
Brief Title: Safety and Efficacy of Ustekinumab in Patients With Palmo-Plantar Pustular Psoriasis or With Palmo-Plantar Pustulosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Manufacturer ceased to produce vials used for this study.
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Janssen-Ortho LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inno-6012
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Palmo-Plantar Pustular Psoriasis; Palmo-Plantar Pustulosis
Keywords: Ustekinumab, Palmo-Plantar, Pustular Psoriasis, Pustulosis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ustekinumab (Active Comparator): Ustekinumab S/C 45mg or 90mg depending on patient's weight or placebo injection. 10 with PPPP and 10 with PPP will receive ustekinumab at Day 0, Weeks 4 and 16 and placebo at Week 20
  Interventions: Drug: Ustekinumab
- Placebo (Placebo Comparator): Placebo S/C (Sodium Chloride). 10 with PPPP and 10 with PPP will receive placebo at Weeks 0 and 4 and ustekinumab at Weeks 16 and 20
  Interventions: Drug: Placebo (Soduim Chloride)

INTERVENTIONS:
Drug: Ustekinumab — Patients randomized to ustekinumab (10 with PPPP and 10 with PPP) will receive ustekinumab at Day 0, Weeks 4 and 16 and placebo at Week 20
  Arms: Ustekinumab
Drug: Placebo (Soduim Chloride) — Patients randomized to placebo (10 with PPPP and 10 with PPP) will receive placebo at Weeks 0 and 4 and ustekinumab at Weeks 16 and 20
  Arms: Placebo

SUMMARY:
This study will provide data on sasety and efficacy of Ustekinumab in patients suffering from Palmo-Plantar Pustular Psoriasis (PPPP) or Palmo-Plantar Pustulosis(PPP)

DETAILED DESCRIPTION:
Twenty patients with active Palmo-Plantar Pustular Psoriasis (cohort A) and twenty patients with active Palmo-Plantar Pustulosis (cohort B) will be included in this placebo-controlled double-blind study.Patients in each cohort will be randomized (1:1) to receive either ustekinumab S/C (Sub-Cutaneous) (45 mg for patients weighting 100 kg or less, and 90 mg for patients weighting more than 100 kg) or placebo.

Patients randomized to ustekinumab (10 with PPPP and 10 with PPP) will receive ustekinumab at Day 0, Weeks 4 and 16 and placebo at Week 20 whereas patients randomized to placebo (10 with PPPP and 10 with PPP) will receive placebo at Weeks 0 and 4 and ustekinumab at Weeks 16 and 20.

Patients will be seen at screening, Day 0, Weeks 4, 8, 16, 20, 24 and 28. The PPPASI (Palmo-Plantar Pustular Area and Severity Index), PPPGA (Palmo-Plantar Physician Global Assessment), PPSA (Palmo-Plantar Surface Area) will be used to evaluate severity and DLQI (Dermatology Life Quality Index), WPAI:PSO (Work Productivity and Activity Impairement Questionnaire:Psoriasis) and PPQoLI (Palmo-Plantar Quality of Life Index)will be used to evaluate quality of life. Safety will be assessed by physical examinations, evaluation of adverse events and laboratory analyses.

High quality digital medical photographs of palms and soles will be taken at Day 0, Weeks 4, 16 and 28. In addition, one optional skin biopsy from a palm or a sole will be performed at Day 0 and Week 16 and pus will be collected from pustules on palms and/or soles at Day 0 and Week 16. Finally, blood will be collected at Day 0 for genetic analysis from every patient who consents to DNA blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* Have had for at least 6 months either:

  * Palmo-plantar pustular psoriasis defined as active palmo-plantar disease morphology suggestive of psoriasis with at least one plaque of typical psoriasis outside the palms and soles or a history of typical plaque psoriasis outside the palms and soles (cohort A) OR
  * Palmo-plantar pustulosis defined as active palmo-plantar morphology suggestive of palmo-plantar pustulosis without lesions of psoriasis outside palms and soles and without a history of psoriasis (cohort B).
* PPPASI score of at least 8 on hands and/or feet and a PPPGA score of 3 (moderate) or 4 (severe) at Day 0
* Stable palmo-plantar pustular psoriasis or palmo-plantar pustulosis for the past 4 weeks
* Men or women 18 years of age or older at time of consent
* Must be candidate for phototherapy and systemic therapy
* Unless surgically sterile (or at least 1 year post-menopausal for women), or abstinent, patient (male or female) is willing to use an effective method of contraception for at least 30 days before Day 0 and until at least 12 months after the last drug administration. Effective method of contraception are:

  * Condom with spermicide, sponge with spermicide, foams with spermicide, jellies with spermicide, diaphragm with spermicide
  * Intra uterine device (IUD)
  * Contraceptives (oral or parenteral)
  * Nuvaring
  * Vasectomy or vasectomised partner
  * Surgically sterile or post-menopausal partner
  * Same-sex partner
* Capable of giving informed consent and the consent must be obtained prior to any study related procedures
* Are considered eligible according to the following TB (Tuberculosis) screening criteria:

  * Have no history of latent or active TB prior to screening Patients with latent TB discovered at screening are not eligible for this study, even if they receive isoniazide or rifampin prophylaxis.
  * No signs or symptoms suggestive of active TB upon medical history and/or physical examination.
  * No recent close contact with a person with active TB or, if there was such contact, have a negative QuantiFERON-TB Gold test (or a negative tuberculin (less than 5mm) skin test when QuantiFERON-TB Gold is not available) and have been referred to a physician specializing in TB to undergo additional evaluation to rule out TB infection.
  * Within 6 weeks prior to the first administration of study agent, have a negative QuantiFERON-TB Gold test. For patients enrolled at sites that where QuantiFERON-TB Gold test is not available, have a negative tuberculin (less than 5mm) skin test.
  * A chest radiograph (posterior-anterior as defined by site-specific requirements), taken within 3 months prior to the first administration of study agent and read by a qualified radiologist, with no evidence of current active TB or old inactive TB
* Female patients of childbearing potential have had a negative serum pregnancy test at the screening visit

Exclusion Criteria:

* Have used topical steroids, topical tar preparations or other topical anti-psoriatic preparations within 2 weeks preceding Day 0 except for the following which is allowed- mild to moderate potency topical corticosteroids for the face, groin, axilla, genitalia and scalp as long as they are applied with gloves: hydrocortisone, desonide, hydrocortisone valerate
* Have presence of erythrodermic or generalized pustular psoriasis
* Have presence of acute forms of tinea pedis and other causes of pustular eruptions of palms and soles apart from PPPP or PPP based on clinical evaluation or evidence of any skin condition that would interfere with the evaluation of PPPP or PPP
* Have had, based on investigator's judgment, any significant infection within 30 days preceding Day 0
* Have used any investigational drugs within 4 weeks of Day 0 or 5 times the half-life of the investigational agent prior to the first administration of study agent, whichever is longer
* Have used systemic anti-psoriatic drugs such as steroids, retinoids, cyclosporine, or methotrexate within 4 weeks of Day 0
* Have used any biologic such as alefacept, etanercept, adalimumab or infliximab within 12 weeks or 5 half-lives which ever is longer of Day 0
* Have received ultraviolet light therapy: UVB (Ultraviolet B), nbUVB (Narrow Band Ultraviolet B), PUVA (Psoralen Ultraviolet A), or tanning bed within 4 weeks of Day 0
* Have had any severe, progressive or uncontrolled renal, hepatic, endocrine, cardiac, gastrointestinal, pulmonary, neurologic, psychiatric, cerebral, hematologic medical condition
* Are known to be infected with hepatitis B, hepatitis C virus or Human Immunodeficiency Virus (HIV)
* Are currently treated for latent tuberculosis
* Have or have had a serious infection (eg: sepsis, pneumonia or pyelonephritis) or have been hospitalized or received IV (Intravenous) antibiotics for an infection during the 2 months prior to screening
* Have any known malignancy or have a history of malignancy (with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to the first administration of study agent)
* Have received within 3 months (within 1 year for BCG (Bacillus Calmette-Guérin) vaccination) prior to the first injection a live virus or bacterial vaccination. Patients must agree not to receive a live virus or bacterial vaccination during the trial or up to 12 months after the last study agent injection
* Have a clinically significant laboratory result that, in the opinion of the investigator, prevents ustekinumab administration for safety reasons
* Are pregnant, nursing or planning pregnancy (both men and women) while enrolled in the study
* Are known to have had a substance abuse (drug or alcohol) problem within the previous 12 months
* Have known hypersensitivity to ustekinumab or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with PPPP who reach PPPASI-50 at Week 16 for patients randomized to ustekinumab as compared to patients randomized to placebo | 16 week
Proportion of patients with PPP who reach PPPASI-50 at Week 16 for patients randomized to ustekinumab as compared to patients randomized to placebo. | 16 Weeks

SECONDARY OUTCOMES:
Evaluation of safety of ustekinumab as compared to placebo by reporting the incidence rates of adverse events and serious adverse events in patient with PPPP | 28 Weeks
Proportion of patients with PPPP who reach PPPASI-75 at Week 16 for patients randomized to ustekinumab as compared to patients randomized to placebo | 16 Weeks
Changes from baseline in PPPASI at Week 16 for patients with PPPP randomized to ustekinumab as compared to patients randomized to placebo | baseline to 16 Weeks
Changes from baseline in the PPPGA at Week 16 for patients with PPPP randomized to ustekinumab as compared to patients randomized to placebo | baseline to 16 Weeks
Changes from baseline in PPSA at Week 16 for patients with PPPP randomized to ustekinumab as compared to patients randomized to placebo | baseline to 16 Weeks
Changes from baseline in the DLQI at Week 16 for patients with PPPP randomized to ustekinumab as compared to patients randomized to placebo | baseline to 16 Weeks
Changes from baseline in WPAI:PSO at Week 16 for patients with PPPP randomized to ustekinumab as compared to patients randomized to placebo | baseline to 16 weeks
Changes from baseline in PPQoLI at Week 16 for patients with PPPP randomized to ustekinumab as compared to patients randomized to placebo | baseline to 16 Weeks
Changes from baseline in PPPP at Week 28 for patients randomized to ustekinumab as measured with the PPPASI, PPPGA, PPSA, DLQI, WPAI:PSO and PPQoLI. | baseline to 28 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Simon Nigen, MD, Principal Investigator — Innovaderm Research Inc.
Locations (8):
- Canada (8):
  - Kirk Barber Research, Calgary, Alberta
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates Ltd, Halifax, Nova Scotia
  - Lynderm Research, Markham, Ontario
  - Windsor Clinical Research Inc., Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherches Dermatologiques du Quebec Metropolitain, Québec, Quebec
  - Clinique Médicale Dr Isabelle Delorme, Saint-Hyacinthe, Quebec